CLINICAL TRIAL: NCT05494294
Title: Does the De-epithelialization Procedure Affect the Epithelial Remnants and Recession Coverage Outcomes?
Brief Title: Comparison of Different De-epithelialization Techniques of Soft Tissue Grafts.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gencay Keceli, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: quality of graft
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Connective Tissue Graft Harvesting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients were randomly assigned into intraorally de-epithelialization group (n=25) and extraorally de-epithelialization group (n=25) groups by one of the authors with an allocation ratio of 1:1 using a computer-generated program after successful completion of the phase I periodontal treatment. One calibrated author masked the applied surgical technique and recorded all clinical variables. The surgeon opened the labeled envelope containing the intervention name.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral (Active Comparator): In this group, the grafts were de-epithelialized at the donor site before harvesting. The calibrated surgeon removed the epithelium with a sharp Kirkland knife under magnification. To be sure of the elimination whole epithelial layer, bleeding was observed. Recipient site was prepared as follows; A after sulculer incision had done (blade 15c) two vertical incions were made from the gingival margin to 3 mm beyond the mucogingival junction A partial-thickness flap was elevated under the recession area and full thickness flap elevated adjacent flap portions. then relasing incisions were made apically from the mucogingival junction. After the preparation of the recipient site, obtained graft was sutured 1 mm apically to the cemento-enamel junction. Finally flap was positioned without tension and stabilized at least 2mm coronally from the cemento-enamel margin with the single interrupted sutures.
  Interventions: Procedure: Intraorally de-epithelialization
- Extraoral (Active Comparator): In this group, the grafts were de-epithelialized after graft harvesting. The calibrated surgeon removed the epithelium with 15 c knife under magnification. all remnants were removed under magnification. Same recipient site procedure was conducted in this group.
  Interventions: Procedure: Extraorally de-epithelialization

INTERVENTIONS:
Procedure: Intraorally de-epithelialization — In this group, the grafts were de-epithelialized at the donor site before harvesting. The calibrated surgeon removed the epithelium with a sharp Kirkland knife under magnification. To be sure of the elimination whole epithelial layer, bleeding was observed. Recipient site was prepared as follows; A after sulculer incision had done (blade 15c) two vertical incions were made from the gingival margin to 3 mm beyond the mucogingival junction A partial-thickness flap was elevated under the recession area and full thickness flap elevated adjacent flap portions. then relasing incisions were made apically from the mucogingival junction. After the preparation of the recipient site, obtained graft was sutured 1 mm apically to the cemento-enamel junction. Finally flap was positioned without tension and stabilized at least 2mm coronally from the cemento-enamel margin with the single interrupted sutures.
  Arms: Intraoral
Procedure: Extraorally de-epithelialization — In this group, the grafts were de-epithelialized after graft harvesting. The calibrated surgeon removed the epithelium with 15 c knife under magnification. all remnants were removed under magnification. Same recipient site procedure was conducted in this group.
  Arms: Extraoral

SUMMARY:
In this randomized comparative controlled clinical trial, 50 patients with single recession defects with thin phenotype were treated with coronally advanced flap. The connective tissue graft was obtained by removing the keratinized layer of the tissue. Removal of the epithelium was achieved by to different approach. At first group epithelium and remnants were removed extraorally whereas others were intraorally. After the removal, obtained graft laid on a lamella, and residual keratinocytes were observed under the microscope. Amount of recession reduction recorded at the 6th week, 6th month, 12th month, and keratinized tissue height, gingival thickness, recession depth, recession width, probing depth, and clinical attachment level, were also evaluated. Keratinized tissue change, Gingival thickness change, root coverage, clinical attachment gain, and complete root coverage were calculated. Wound healing index, tissue appearance, patient expectations, aesthetics, and dentine hypersensitivity were assessed at baseline and 6th week.

ELIGIBILITY:
Inclusion Criteria:

* Single tooth recession more than 2mm
* Gingival thickness less than 1mm

Exclusion Criteria:

* unstable endodontic conditions or presence of any restoration/abrasion,
* tooth mobility, any surgical history or gingival enlargement in the area,
* smoking
* uncontrolled systemic disease, pregnancy or use of drugs known to affect gingival conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Recession reduction | 3rd month
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession reduction | 6th month
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession reduction | 12th month
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.

SECONDARY OUTCOMES:
amount of deciduous cells | at the day of the surgery.
  Amount of deciduous cells was measured with computerized microscope via histomorfometric methods.
percentage of deciduous cells | at the day of the surgery
  amount of deciduous cells Amount of deciduous cells was measured with computerized microscope via histomorfometric methods.
Recession Depth (RD) | Baseline.
  RD, was measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession Depth (RD) | 3rd month
  RD, was measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession Depth (RD) | 6th month
  RD, was measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession Depth (RD) | 12th month
  RD, was measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Keratinized Tissue Height (KTH) | baseline
  TH, was measured from gingival margin to the mucogingival junction (MGJ).
Keratinized Tissue Height (KTH) | 3rd month
  TH, was measured from gingival margin to the mucogingival junction (MGJ).
Keratinized Tissue Height (KTH) | 6th month
  TH, was measured from gingival margin to the mucogingival junction (MGJ).
Keratinized Tissue Height (KTH) | 12th month
  TH, was measured from gingival margin to the mucogingival junction (MGJ).
Gingival Thickness (GT) | baseline
  GT, was measured at the midpoint location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Gingival Thickness (GT) | 3rd month
  GT, was measured at the midpoint location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Gingival Thickness (GT) | 6th month
  GT, was measured at the midpoint location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Gingival Thickness (GT) | 12th month
  GT, was measured at the midpoint location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Recession width (RW) | baseline
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Recession width (RW) | 3rd month
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Recession width (RW) | 6th month
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Recession width (RW) | 12th month
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Probing pocket depth (PD) | baseline
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Probing pocket depth (PD) | 3rd month
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Probing pocket depth (PD) | 6th month
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Probing pocket depth (PD) | 12th month
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | Baseline
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | 3rd month
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | 6th month
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | 12th month
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Keratinized tissue change (KTC) | 3rd month
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Keratinized tissue change (KTC) | 6th month
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Keratinized tissue change (KTC) | 12th month
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Wound healing index (WHI) | 3rd month
  Wound healing index (WHI) was recorded two-weeks after surgery. The wound surface was visually inspected and the soft tissue healing was defined as 'uneventful' (score 1), 'slightly disturbed' (score 2) or 'poor' (score 3) based on the presence and severity of the items including patient discomfort, erythema, edema, suppuration and flap dehiscence.
Wound healing index (WHI) | 6th month
  Wound healing index (WHI) was recorded two-weeks after surgery. The wound surface was visually inspected and the soft tissue healing was defined as 'uneventful' (score 1), 'slightly disturbed' (score 2) or 'poor' (score 3) based on the presence and severity of the items including patient discomfort, erythema, edema, suppuration and flap dehiscence.
Wound healing index (WHI) | 12th month
  Wound healing index (WHI) was recorded two-weeks after surgery. The wound surface was visually inspected and the soft tissue healing was defined as 'uneventful' (score 1), 'slightly disturbed' (score 2) or 'poor' (score 3) based on the presence and severity of the items including patient discomfort, erythema, edema, suppuration and flap dehiscence.
Tissue appearance (TA) | 3rd month
  Tissue appearance (TA) was evaluated by asking the patients to score the consistency, contour, color match, keloid formation degree and contiguity of their treated sites at T2. The scores were collected as points, shown in parentheses, by asking the consistency as firm (1p) or spongy (0p); contour as presence (2p) or absence (0p) of knife-edged and scalloped gingival margin; color match as excellent (3p), good (2p), adequate (1p) or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); contiguity as the presence (-1p) or absence (0p) of each perceptible incision mark.
Tissue appearance (TA) | 6th month
  Tissue appearance (TA) was evaluated by asking the patients to score the consistency, contour, color match, keloid formation degree and contiguity of their treated sites at T2. The scores were collected as points, shown in parentheses, by asking the consistency as firm (1p) or spongy (0p); contour as presence (2p) or absence (0p) of knife-edged and scalloped gingival margin; color match as excellent (3p), good (2p), adequate (1p) or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); contiguity as the presence (-1p) or absence (0p) of each perceptible incision mark.
Tissue appearance (TA) | 12th month
  Tissue appearance (TA) was evaluated by asking the patients to score the consistency, contour, color match, keloid formation degree and contiguity of their treated sites at T2. The scores were collected as points, shown in parentheses, by asking the consistency as firm (1p) or spongy (0p); contour as presence (2p) or absence (0p) of knife-edged and scalloped gingival margin; color match as excellent (3p), good (2p), adequate (1p) or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); contiguity as the presence (-1p) or absence (0p) of each perceptible incision mark.
Dentine hypersensitivity (DH) | 3rd month
  Dentine hypersensitivity (DH) was evaluated with air evaporative stimulus method at baseline and T2. After placement of finger(s) for preserving the nearby teeth, the recession sites were subjected to evaporative stimulus comprised of 1-second air blast from 1 to 3 mm distance by using the air spray at 40-65 psi pressure and 19±50C. After application, the patients were requested to give a score to their DH between 0 (=no pain) and 10 (=extreme pain).
Dentine hypersensitivity (DH) | 6th month
  Dentine hypersensitivity (DH) was evaluated with air evaporative stimulus method at baseline and T2. After placement of finger(s) for preserving the nearby teeth, the recession sites were subjected to evaporative stimulus comprised of 1-second air blast from 1 to 3 mm distance by using the air spray at 40-65 psi pressure and 19±50C. After application, the patients were requested to give a score to their DH between 0 (=no pain) and 10 (=extreme pain).
Dentine hypersensitivity (DH) | 12th month
  Dentine hypersensitivity (DH) was evaluated with air evaporative stimulus method at baseline and T2. After placement of finger(s) for preserving the nearby teeth, the recession sites were subjected to evaporative stimulus comprised of 1-second air blast from 1 to 3 mm distance by using the air spray at 40-65 psi pressure and 19±50C. After application, the patients were requested to give a score to their DH between 0 (=no pain) and 10 (=extreme pain).
Aesthetics (A) | 3rd month
  Aesthetics (A) was evaluated by the patient at T1 by rating its level as excellent, good, fair or poor.
Aesthetics (A) | 6th month
  Aesthetics (A) was evaluated by the patient at T1 by rating its level as excellent, good, fair or poor.
Aesthetics (A) | 12th month
  Aesthetics (A) was evaluated by the patient at T1 by rating its level as excellent, good, fair or poor.
Vestibuler Depth | baseline
  VD was measured from the gingival margin to the deepest point of to vestibule sulcus.
Vestibuler Depth | 3rd month
  VD was measured from the gingival margin to the deepest point of to vestibule sulcus.
Vestibuler Depth | 6th month
  VD was measured from the gingival margin to the deepest point of to vestibule sulcus.
Vestibuler Depth | 12th month
  VD was measured from the gingival margin to the deepest point of to vestibule sulcus.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Din F, Kabalak MO, Yilmaz BT, Baris E, Avci H, Caglayan F, Keceli HG. Efficacy of different gingival graft de-epithelialization methods: A parallel-group randomized clinical trial. Clin Oral Investig. 2025 May 7;29(6):289. doi: 10.1007/s00784-025-06365-7. PMID 40332625